CLINICAL TRIAL: NCT03470311
Title: Benralizumab in Patients With Inadequate Response to Anti-IL5 Monoclonal Antibody Therapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-12992
Record Dates: First submitted 2018-03-01; First posted 2018-03-19 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Severe Prednisone Dependent Eosinophilic Asthma
Keywords: Eosinophils; asthma; inflammation; prednisone
MeSH Terms: conditions — Asthma; Inflammation | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Benralizumab (Active Comparator): Benralizumab 30mg in 1mL subcutaneously
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Matched placebo (1mL) to active Benralizumab subcutaneously
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — 30mg in 1mL pre-filled syringe
  Other Names: MEDI-563
  Arms: Benralizumab
Biological: Placebo — Matched placebo (1mL) in pre-filled syringe
  Arms: Placebo

SUMMARY:
In severe prednisone-dependent eosinophilic asthma, Benralizumab would suppress airway eosinophilia that is not suppressed by either Mepolizumab or Reslizumab and this would be associated with greater asthma control

DETAILED DESCRIPTION:
Benralizumab thus targets 'eosinophil biology', by inhibiting the interleukin (IL-5) receptor signalling, and inducing apoptosis in cells with an IL-5receptor. Hence, for patients who remain 'uncontrolled' on anti-IL-5 therapy (with detectable eosinophil activity and IL5-Rα+ cells in the airways), the investigators believe would benefit from a strategy that not only reduces eosinophil proliferation/recruitment/maturation, but also depletes cells capable of inducing downstream IL-5 signalling.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent Prior to the beginning of the study, patients must be willing and fully capable to provide written informed consent.
2. Diagnosed prednisone-dependent eosinophilic asthma
3. Previous treatment with 100 mg mepolizumab administered subcutaneously Q4W or reslizumab 3 mg/kg IV Q4W for at least 6 months
4. Sputum eosinophils >3%
5. ACQ ≥1.5
6. Age >18
7. Male or eligible female subjects:

   To be eligible for entry into the study, females of childbearing potential (premenopausal women who are not permanently sterilized by means of hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) must commit to consistent and correct use of a highly effective method of birth control (true sexual abstinence, a vasectomized sexual partner, Implanon, female tubal occlusion, Intrauterine device (IUD), Depo provera injections, oral contraceptive pills or Nuvaring) for the duration of the trial and for 3 months after the last study drug administration. A serum pregnancy test is required of all females at the initial Baseline Visit (Visit 1). In addition, a urine pregnancy test will be performed for all females prior to enrollment, during each scheduled study visit prior to the injection of investigational product, and during the Follow-up Visit.
8. Male subjects who are sexually active must agree to use a double barrier method of contraception (condom with spermicide) from the first dose of study drug and for 3 months after the last dose of study drug.

Exclusion Criteria:

1. Currently receiving another monoclonal antibody
2. Intolerance, hypersensitivity, insensitivity or neutralizing antibody to Mepolizumab and/or Reslizumab
3. Malignancy within the last 5 years
4. Any co-morbidity that the investigator believes is a contraindication. This includes but is not limited to any respiratory, cardiovascular, gastrointestinal, hematological, neurological, immunological, musculoskeletal, renal, infectious, neoplastic or inflammatory condition that may place the safety of the subject at risk during the duration of the study, influence the results of the study or their interpretation, or prevent the patient from completing the entire duration of the study.
5. Current pregnancy or lactation
6. Current smoker or ex-smoker with a smoking history greater than 20 pack years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Sputum eosinophil percentage | Visit 1 (Week 2) and Visit 10 (Week 38)
  Change in Percentage of sputum eosinophils (%)

SECONDARY OUTCOMES:
Blood eosinophils | Visit 1 (Week 2) and Visit 10 (Week 38)
  Blood eosinophil level (x10^9/L)
Forced Expired Volume in 1 second (FEV1)(pre and post bronchodilator) | Visit 1 (Week 2) and Visit 10 (Week 38)
  FEV1 in litres both pre and post bronchodilator
ACQ-5 (Asthma Control Questionnaire) | Visit 1 (Week 2) and Visit 10 (Week 38)
  Asthma Control Questionnaire score (mean answer of 5 questions on a 7-point scale (0=no impairment, 6= maximum impairment).
Fraction of exhaled nitric oxide (FeNO) | Visit 1 (Week 2) and Visit 10 (Week 38)
  Exhaled nitric oxide measurement in ppb
Number of Exacerbations (defined as: ER visit/hospitalization requiring prednisone burst) | Visit 1 (Week 2) and Visit 10 (Week 38)
  Worsening requiring increase in oral steroids/prednisone (30mg x 5 days)
Sputum and blood ILC2 biology | Visit 1 (Week 2) and Visit 10 (Week 38)
  Measurement of ILC2 biological cells in both blood and sputum
Sputum autoimmune responses | Visit 1 (Week 2) and Visit 10 (Week 38)
  Measurement of autoimmune markers in sputum: anti-eosinophil peroxidase (EPX) and anti-nuclear antibodies (ANA) - (See last reference PubMed ID: 28751233)

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD, PhD, Principal Investigator — McMaster University and St. Joseph's Healthcare Hamilton
Locations (1):
- Firestone Institute for Respiratory Health, Research - St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mukherjee M, Lim HF, Thomas S, Miller D, Kjarsgaard M, Tan B, Sehmi R, Khalidi N, Nair P. Airway autoimmune responses in severe eosinophilic asthma following low-dose Mepolizumab therapy. Allergy Asthma Clin Immunol. 2017 Jan 6;13:2. doi: 10.1186/s13223-016-0174-5. eCollection 2017. PMID 28070196
- [Background] Smith SG, Chen R, Kjarsgaard M, Huang C, Oliveria JP, O'Byrne PM, Gauvreau GM, Boulet LP, Lemiere C, Martin J, Nair P, Sehmi R. Increased numbers of activated group 2 innate lymphoid cells in the airways of patients with severe asthma and persistent airway eosinophilia. J Allergy Clin Immunol. 2016 Jan;137(1):75-86.e8. doi: 10.1016/j.jaci.2015.05.037. Epub 2015 Jul 17. PMID 26194544
- [Background] Sehmi R, Smith SG, Kjarsgaard M, Radford K, Boulet LP, Lemiere C, Prazma CM, Ortega H, Martin JG, Nair P. Role of local eosinophilopoietic processes in the development of airway eosinophilia in prednisone-dependent severe asthma. Clin Exp Allergy. 2016 Jun;46(6):793-802. doi: 10.1111/cea.12695. PMID 26685004
- [Background] Kolbeck R, Kozhich A, Koike M, Peng L, Andersson CK, Damschroder MM, Reed JL, Woods R, Dall'acqua WW, Stephens GL, Erjefalt JS, Bjermer L, Humbles AA, Gossage D, Wu H, Kiener PA, Spitalny GL, Mackay CR, Molfino NA, Coyle AJ. MEDI-563, a humanized anti-IL-5 receptor alpha mAb with enhanced antibody-dependent cell-mediated cytotoxicity function. J Allergy Clin Immunol. 2010 Jun;125(6):1344-1353.e2. doi: 10.1016/j.jaci.2010.04.004. PMID 20513525
- [Background] Mukherjee M, Aleman Paramo F, Kjarsgaard M, Salter B, Nair G, LaVigne N, Radford K, Sehmi R, Nair P. Weight-adjusted Intravenous Reslizumab in Severe Asthma with Inadequate Response to Fixed-Dose Subcutaneous Mepolizumab. Am J Respir Crit Care Med. 2018 Jan 1;197(1):38-46. doi: 10.1164/rccm.201707-1323OC. PMID 28915080
- [Background] Nair P, Wenzel S, Rabe KF, Bourdin A, Lugogo NL, Kuna P, Barker P, Sproule S, Ponnarambil S, Goldman M; ZONDA Trial Investigators. Oral Glucocorticoid-Sparing Effect of Benralizumab in Severe Asthma. N Engl J Med. 2017 Jun 22;376(25):2448-2458. doi: 10.1056/NEJMoa1703501. Epub 2017 May 22. PMID 28530840
- [Background] Mukherjee M, Bulir DC, Radford K, Kjarsgaard M, Huang CM, Jacobsen EA, Ochkur SI, Catuneanu A, Lamothe-Kipnes H, Mahony J, Lee JJ, Lacy P, Nair PK. Sputum autoantibodies in patients with severe eosinophilic asthma. J Allergy Clin Immunol. 2018 Apr;141(4):1269-1279. doi: 10.1016/j.jaci.2017.06.033. Epub 2017 Jul 24. PMID 28751233